CLINICAL TRIAL: NCT00067379
Title: Early Orthodontic Intervention Under Medicaid
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Northwest and Alaska Center on Oral Health Disparities (Other); Washington State Department of Social and Health Services (Other); Seattle Children's Hospital (Other)
Responsible Party: Gregory King, DMD, PhD, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIDCR-142542; U54DE014254 (NIH)
Record Dates: First submitted 2003-08-15; First posted 2003-08-19 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Medicaid patients with medically necessary malocclusions treated during the mixed dentition with limited goals followed by observation
  Interventions: Procedure: interceptive orthodontic treatments

INTERVENTIONS:
Procedure: interceptive orthodontic treatments — orthodontic procedures

SUMMARY:
The primary objective of this study is to examine the usefulness of early orthodontic intervention as a means of increasing access to orthodontic services for children of low-income families.

DETAILED DESCRIPTION:
Orthodontic treatment has become a widely accepted procedure in dentistry. The benefits include improved oral health, function, esthetics and quality of life. Significant disparities exist among income strata regarding access to orthodontic services. The sources of these disparities are complex and may reflect differences in the disease prevalence, gender, cultural biases, perception of problems by this population, economic imperatives and negative perceptions of these patients by orthodontists. The primary objective of this study is to examine the usefulness of early orthodontic intervention as a means of increasing access to orthodontic services for children of low-income families.

Aim 1. To compare orthodontic outcomes, facial body image, and quality of life between Medicaid participants who receive early orthodontic treatment and those who do not. 1.a To compare the level of understanding and compliance between early treatment subjects given information about the goals, risks and benefits of the planned treatment one-on-one by an orthodontist, with subjects who also use an interactive CD-ROM to provide this information. This will be referred to as the Informed Consent Study and should not be confused with the routine informed consenting process used to enroll subjects into the overall study.Aim 2. To compare orthodontic outcomes, facial body image, and quality of life between Medicaid-funded and private-pay patients who receive full orthodontic treatment at adolescence.Aim 3. To compare orthodontic outcomes, facial body image, and quality of life between Medicaid-funded patients who receive early orthodontic treatment only and Medicaid-funded participants who receive full orthodontic treatment at adolescence. Relationship of this project with the Disparity Center theme. Two of the goals of the Northwest and Alaska Center for Oral Health Disparity are met by this study. The first is to conduct clinical research to evaluate the efficacy of interventions to prevent and treat oral diseases and conditions in children. The second is to develop community-based research that translates existing knowledge and new information regarding children and their caretakers into new technologies and interventions that hold promise for reducing disparities. Today, children of low-income families have very limited access to orthodontic treatment. We also know that some relatively simple interventions done during the mixed dentition can be effective at reducing the severity of malocclusion. This study is designed to examine how effective these early orthodontic interventions are in a Medicaid population. It will also examine how outcomes from early treatment in Medicaid patients compare to the more complex approach of complete orthodontic treatment in the permanent dentition. Many orthodontists perceive that Medicaid patients are at risk for poor outcomes, and limit access as a consequence. The follow-up component of this study will address this issue by making a comparison between Medicaid and private-pay patients treated in similar environments. We expect that significantly greater access to orthodontic services could be provided for Medicaid patients by the more widespread use of simpler, more timely interventions. This study will provide data on the trade-off between simple, timely partial treatments, versus complete full treatments. In response to the second theme of the Disparity Center, the use of interactive CD-ROMs that provide treatment information at the comprehension level of young patients and their parents, and in a culturally appropriate manner, will be examined. We expect this approach will improve patient and parent understanding of the proposed treatment, as well as enhancing compliance with treatment procedures in order to assure successful outcomes.

ELIGIBILITY:
"Inclusion Criteria:"

* Enrolled in Medicaid
* Fluency in English, Spanish, Vietnamese, Chinese, Somalian or Ethiopian
* Acceptable malocclusion
* Free of oral disease
* Current immunizations and record of dental care
* Acceptable oral hygiene
* Anticipate living in the area for 4 years
* Absence of craniofacial anomalies
* Absence of unilateral posterior crossbite with facial asymmetry
* No prior orthodontic treatment
* Agree to be randomized to early orthodontic treatment or late full treatment
* Signs assent/consent

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2003-04; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Peer Assessment Rating | Pre-study, post - early treatment or observation, post full treatment or observation

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J King, DDS, Principal Investigator — University of Washington
Locations (1):
- Odessa Brown Children's Clinic, Seattle, Washington, United States

REFERENCES:
- [Derived] King GJ, Spiekerman CF, Greenlee GM, Huang GJ. Randomized clinical trial of interceptive and comprehensive orthodontics. J Dent Res. 2012 Jul;91(7 Suppl):59S-64S. doi: 10.1177/0022034512448663. PMID 22699670